CLINICAL TRIAL: NCT03597919
Title: A Study of Immunogenicity and Seroconversion With Sabin Inactivated Polio Vaccine Schedules in China.
Brief Title: A Study of Immunogenicity and Seroconversion With Sabin IPV Schedules in China.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention, China (Other Government)
Collaborators: Shandong Province Centers for Disease Control and Prevention (Other); World Health Organization (Other)
Responsible Party: Principal Investigator, AN Zhijie, Director of Vaccine Evaluation Division, National Immunization Program, Centers for Disease Control and Prevention, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201717
Record Dates: First submitted 2018-05-23; First posted 2018-07-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Poliomyelitis
Keywords: Inactivated Poliovirus Vaccine; Sabin strain
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Intervention Model Description: a multi-center, randomized, open-label, seroconversion/immunogenicity study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three-dose schedule for Sabin IPV (Active Comparator): Subjects vaccinate Sabin IPV at 2, 3, and 4 months of age,will be collected blood specimens twice - right before the first dose of IPV, and one month after the 3rd dose of IPV.
  Interventions: Biological: Sabin IPV
- Two-dose schedule for Sabin IPV (Experimental): Subjects vaccinate first dose IPV at 4 months, and the second dose IPV given between 8 and 11 months of age,will be collected blood specimens twice - right before the first dose of IPV, and one month after the 2nd dose of IPV.
  Interventions: Biological: Sabin IPV

INTERVENTIONS:
Biological: Sabin IPV — We select one Sabin IPV product, produced by Kunming Bio institute, which is available for China's National Immunization Program in the selected study sites.
  Other Names: Sabin strain Inactivated Poliovirus Vaccine

SUMMARY:
In April 2017, WHO recommended that a two-dose, Inactivated Poliovirus Vaccine, IPV-only schedule at 4 months and 8 months of age can be used after polio eradication, with a schedule seroconversion target of at least 90%. However, there is no such data for China domestic Sabin strain IPVs to support a 2-dose schedule among Chinese infants.

This research is to determine the seroconversion rates among two arms:

Group 1: two-dose schedule, infants will be received two doses of Sabin IPV, the first dose at 4 month of age, and the second dose at 8-11 month of age.

Group 2: three-dose schedule, infants will be received three doses of Sabin IPV at 2, 3 and 4 month of age respectively. This schedule is currently recommended by manufacture's package insert for routine use.

The hypothesis is the seroconversion will be above 90% in both groups.

DETAILED DESCRIPTION:
As a part of global polio eradication endgame immunization strategy, WHO requested all OPV-using countries to introduce at least one dose of IPV into the routine immunization schedule. Ideally IPV should be administered after 14 weeks of age, however an IPV-OPV sequential schedule is acceptable if VAPP is a concern. China stopped trivalent OPV in routine immunization in May 2016, introduced one dose of IPV at 2 months followed by three doses of type I / III bivalent OPV (bOPV) at 3 and 4 months and 4 years. A Sabin strain IPV was licensed in January 2015, and a second Sabin IPV was approved by China FDA in September 2017. The production capacity will increase in the next few years and will meet the demands of an IPV-only schedule in China. Other Sabin IPVs are in clinical trial stages, which will lead to sufficient IPV production for China to export IPV.

In April 2017, WHO/SAGE recommended that a two-dose, IPV-only schedule can be used after polio eradication, with a schedule seroconversion target of at least 90%. The recommendation was based in part on a study conducted in Cuba using Salk-IPV at 4 months and 8 months of age. Considering that risk of polio virus transmission is decreasing over time, and that IPV - either domestic Sabin-IPV or imported Salk-IPV - is expensive (6 USD/dose) for a program serving a birth cohort of 18 million, an efficient two-dose, IPV-only schedule will be very competitive with a more traditional 4-dose IPV-only schedule. However, for domestic Sabin IPVs, there are no such data to support a 2-dose schedule among Chinese infants.

The overall objective of this research is to determine the seroconversion rates of two reduced Sabin IPV schedules in Chinese children - a 2-dose schedule and a 3-dose schedule.

Group 1: two-dose schedule, infants will be received two doses of Sabin IPV, the first dose at 4 month of age, and the second dose at 8-11 month of age.

Group 2: three-dose schedule, infants will be received three doses of Sabin IPV at 2, 3 and 4 month of age respectively. This schedule is currently recommended by manufacture's package insert for routine use.

The hypothesis is the seroconversion will be above 90% in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian agree to participate in our study.
* The family is living locally with legal residency status.

Exclusion Criteria:

* Parent or legal guardian does not agree to participate in our study.
* The potential subject has received IPV or OPV before 4 months of age in the two-dose schedule group.
* The potential subject has one or more contraindications to IPV (although we will note the contraindications).

Ages: 2 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 560 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate | 10 months
  Determine whether the seroconversion rate is above 90% using a two-dose Sabin IPV alone schedule with the first dose Sabin IPV given at 4 months and the second dose Sabin IPV given ≥4 months after the first dose.

SECONDARY OUTCOMES:
Neutralizing antibody titers | 10 months
  Measure neutralizing antibody titers against poliovirus type I, II and III among two-dose Sabin IPV-only schedules compared with three-dose Sabin IPV alone schedule.

CONTACTS AND LOCATIONS:
Overall Officials: Zijian Feng, MD, MPH, Study Chair — Centers for Disease Control and Prevention, China
Locations (1):
- Shandong Center for Disease Control and Prevention, Jinan, China

IPD SHARING:
Plan to Share IPD: No